CLINICAL TRIAL: NCT02969876
Title: Pattern Separation, Brain Derived Neurotrophic Factors, and Mechanisms of Vortioxetine
Acronym: VOR-IISR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Site was unable to reach Sponsor recruitment goals.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Bipolar Clinic and Research Program; Associate Director, Depression Clinical and Research Program; Director, Clinical Research Support Office, Clinical Research Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P001243
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Depressive Disorder; Major Depression; Depression; Depression, Unipolar
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Phase (Other): During this phase participants receive open label vortioxetine for 6 weeks. Participants come to the Depression Clinical & Research Program at the Massachusetts General Hospital for visits once a week. During these visits the participants meet with clinicians and complete cognitive tasks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine is a selective serotonin re-uptake inhibitor (SSRI), a common form of treatment for major depressive disorder.
  Other Names: Trintellix; Brintellix

SUMMARY:
The study is a 6-week, proof-of-concept, open trial of vortioxetine for 20 patients with major depressive disorder.

DETAILED DESCRIPTION:
The U.S. Food and Drug Administration approved vortioxetine to treat major depressive disorder in 2013. Researchers believe vortioxetine may improve pattern separation and pattern completion (i.e., a neurological function) in people with major depressive disorder; thus, this research study aims to determine how vortioxetine increases a person's ability to think. The current study is an open label trial, therefore, all participants will receive vortioxetine. Furthermore, participants receive the vortioxetine at no cost. It will take participants 6 weeks to complete this study. Participants are asked to come to the Mass General Hospital campus for 1 screening visit which includes a full psychiatric evaluation, and 5 additional study visits. During study visits, participants will meet with a clinician and then complete computer based cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

1. Meets Diagnostic and Statistical Manual of Mental Disorders (Versions 4 and 5) criteria for and Major Depressive Disorder.
2. Hamilton Depression Rating Scale-17 score greater than 18.
3. Men and women between ages >=18 and 65.

Exclusion Criteria:

1. Meets Diagnostic and Statistical Manual of Mental Disorders (versions 4 and 5) criteria for schizophrenia, schizoaffective disorder, obsessive compulsive disorder.
2. Unable to follow instructions or otherwise unable to participate in the trial.
3. Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, partner with vasectomy)
4. Patients who, in the investigator's judgment, pose a current, serious suicidal or homicidal risk.
5. Serious or unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease.
6. History of seizure disorder.
7. The following Diagnostic and Statistical Manual of Mental Disorders (Version 4) diagnoses (any current or past history, except substance abuse disorders):

   Organic mental disorders, schizoaffective disorder, delusional disorder, psychotic disorders not elsewhere classified.
8. History of multiple adverse drug reactions or allergy to the study drugs.
9. Patients with mood congruent or mood incongruent psychotic features
10. Current use of other psychotropic drugs.
11. Clinical or laboratory evidence of hypothyroidism.
12. Patients who have failed to respond during the course of their current major depressive episode to at least one adequate antidepressant trial, defined as six weeks or more of treatment with citalopram 40 mg/day (or its antidepressant equivalent)
13. Patients who have had electroconvulsive therapy within the 6 months preceding baseline.
14. Concomitant use of serotonergic agents
15. Meets Diagnostic and Statistical Manual of Mental Disorders (versions 4 and 5) criteria for bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nierenberg, M.D., Principal Investigator — Depression Clinical and Research Program/ Bipolar Clinical and Research Program
Locations (1):
- the Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Trial Vortioxetine: All enrolled participants received open trial of Vortioxetine for 6 weeks.
Period: Overall Study
Arm/Group | Open Trial Vortioxetine
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Phase
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.5 (3.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Quick Inventory of Depressive Symptomatology - Clinician Version (QIDS-C)
Description: This scale is designed to assess the severity of depressive symptoms. The minimum score is a 0 (zero) and the maximum score is a 27, and a higher score means a worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Phase
Number analyzed (Participants) | 2
score on a scale | 12.5 (10.60)

2. Secondary Outcome: Digital Symbol Substitution Test
Description: A cognitive measure sensitive to learning and memory. Participants are given 90 seconds to match as many symbols to numbers according to a key located on the top of the page. A higher score means a better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: number of substitutions
Arm/Group | Open Trial Vortioxetine
Number analyzed (Participants) | 2
number of substitutions | 41.5 (1.5)

3. Secondary Outcome: Rey Auditory Verbal Learning Test
Description: A cognitive measure sensitive to learning and memory. Minimum score is a zero. Maximum score is a 75. A higher score means a better outcome
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: number of words recalled
Arm/Group | Open Trial Vortioxetine
Number analyzed (Participants) | 2
number of words recalled | 54 (1)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Open Trial Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Trial Vortioxetine (N=2)
Tripped, hit knee, went to ER (Musculoskeletal and connective tissue disorders) | 1
Migraines (General disorders) | 1 (1)
Headaches (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT02969876/Prot_SAP_000.pdf